CLINICAL TRIAL: NCT06541067
Title: Study of Posaconazole Prophylaxis in Patients Receiving Hematopoietic Stem Cell Allograft (Allo-HSC) at High Risk of Invasive Fungal Infection (IFI): POSALLO Study
Brief Title: Study of Posaconazole Prophylaxis in Patients Receiving Hematopoietic Stem Cell Allograft (Allo-HSC) at High Risk of Invasive Fungal Infection (IFI)
Acronym: POSALLO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC23_0186
Record Dates: First submitted 2024-07-24; First posted 2024-08-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancy
Keywords: Hematopoietic stem cell allograft (Allo-CSH); Posaconazole; Pharmacology
MeSH Terms: conditions — Hematologic Neoplasms | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Posaconazole (Experimental)
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — Per Os, on Day 0 of allo-CSH if the patient's condition permits, or after the last dose of immunosuppressor (post-transplant cyclophosphamide) (Day+5 or Day+6 depending on protocols).
  On the first day of treatment: 300 mg in the morning (= 3 x 100 mg tablets) and 300 mg in the evening (= 3 x 100 mg tablets), then from day 2 of treatment: 300 mg per day (= 3 x 100 mg tablets) in a single dose

SUMMARY:
Patients receiving an allogeneic hematopoietic stem cell transplant (allo-CSH) are at high risk of infection, particularly of fungal origin. Until the 2018 recommendations of the 6th European Conference on Infections in Leukemia (ECIL6), primary prophylaxis of invasive fungal infections (IFI), in allograft patients, was based on the administration of fluconazole until D100. Due to changes in transplantation practices (alternative donor transplantation, sequential transplantation, etc.) and changes in microbiological ecology (increased incidence of IFIs caused by filamentous germs such as aspergillosis and mycormycosis), fluconazole prophylaxis is now sometimes suboptimal. It is therefore recommended that patients at high risk of developing IFIs should be given azole molecules with activity against filamentous agents as primary prophylaxis during the first 3 months after transplantation.

Posaconazole is often under-dosed (below the minimum effective concentration). It therefore seems essential to carry out a prospective study with close [C]min dosing in the specific situation of allograft patients, a population that appears to be at risk of underdosing in the light of initial retrospective analysis results.

DETAILED DESCRIPTION:
There are several treatments based on azole molecules: voriconazole, posaconazole, isavuconazole... To date, none of these treatments has been approved for primary post-allograft prophylaxis. Posaconazole is indicated in cases of graft-versus-host disease (GVHD) (requiring systemic corticosteroid therapy after allo-CSH), and as primary prophylaxis during aplasia in patients with acute myeloblastic leukemia/myelodysplasia (AML/MDS). Other azole molecules are not approved for primary prophylaxis, and may give rise to drug interactions with certain treatments prescribed for allograft patients (e.g. ciclosporin, letermovir).

Although recommendations for the administration of posaconazole as primary prophylaxis post allo-CSH have been in place for 4 years, few studies are available to date. The adult hematology department of Nantes University Hospital conducted a retrospective study of 70 allograft patients at high risk of IFI between 04/2020 and 12/2021. Posaconazole treatment was administered from D0 (or the day after the 2nd dose of post-transplant cyclophosphamide) to D100. Treatment was generally well tolerated, with discontinuation due to possible treatment toxicity in 12.6% of cases, mainly of hepatic origin (n=7). Posaconazole was resumed in 2 cases without recurrence of toxicity. In 84.2% of patients, no IFI was observed. One of the limitations of this study was the low number of determinations of residual posaconazole concentration ([C]min). In fact, [C]min was carried out in only 59 patients/70, with a median delay of 9 days. In 43% of cases, the [C]min was insufficient (< 0.5 mg/L), which is significantly lower than the [C]min obtained in patients with AML/MDS undergoing induction ([C]min< 0.5 mg/L: 5% of patients). It therefore seems essential to carry out a prospective study with close [C]min measurement in the specific situation of allograft patients, a population that appears to be at risk of underdosing in the light of the initial retrospective results of analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age. There is no maximum age for inclusion
* Allo-CSH transplant for hematologic malignancy or benign hemopathy of any type with one or more high risk IFI criteria:

  * alternative donor (haploidentical intra-family donor, mismatch file donor, placental blood)
  * sequential conditioning for disease not in remission at the time of transplantation
  * use of post-transplant cyclophosphamide (PTCY) for GVH prophylaxis
  * patient who has previously received a HSC allograft
* Written informed consent prior to protocol initiation
* ECOG <=2
* Female of childbearing age with negative pregnancy test and on highly effective contraception during treatment and for 12 months after posaconazole discontinuation
* Men of childbearing age with effective contraception during treatment and for 6 months after stopping posaconazole.
* Hepatitis B, C and HIV serologies negative.
* Social security affiliation

Exclusion Criteria:

* Patients with a history of IFI, whether active or resolved at the time of allografting
* Patient with known intolerance to posaconazole
* Patients with concomitant treatments FORBIDDING association with posaconazole: ergot alkaloids, CYP3A4 substrates (terfenadine, astemizole, cisapride, pimozide, halofantrine or quinidine), HMG-CoA reductase inhibitors (simvastatin, lovastatin and atorvastatin) or any other contraindicated treatment listed in VIDAL
* patients with congenital or acquired QTc prolongation (QTc >470ms)
* Cardiac: systolic ejection fraction < 50% by transthoracic ultrasound or isotopic method (isotopic gamma-angiography)
* Respiratory: DLCOc <40% of theoretical on EFR
* Renal: creatinine clearance < 50 ml/min (assessed using MDRD method)
* Hepatic: transaminases greater than 5 times normal or bilirubin greater than 2 times normal
* Pregnant or breast-feeding women,
* Women or men of childbearing age without effective contraception
* Serious, uncontrolled concomitant infections
* Yellow fever vaccination within the last year
* Patient protected by law (guardianship, curatorship, safeguard of justice)
* Psychological, family, sociological or geographical conditions that may hinder compliance with the study protocol and follow-up schedule
* Patient who does not speak or understand French
* Participation in any other therapeutic study with an exclusion period still in effect at the time of inclusion or planned participation in another therapeutic study while taking posaconazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-11-08 (Estimated)

PRIMARY OUTCOMES:
Effective residual concentration of posaconazole | On the 8th day of treatment (i.e. after 7 days of treatment)
  The main objective is to study, in the early phase after allo-CSH, the percentage of patients who have an effective residual concentration of posaconazole.
  The primary endpoint is plasma residual posaconazole concentration ([C]min), measured on day 8 of posaconazole initiation. A [C]min > 0.7mg/l is considered effective.

SECONDARY OUTCOMES:
Monitoring of residual plasma concentrations [C]min | From posaconazole baseline up to Day100
  Weekly residual plasma concentrations of posaconazole
Description of circumstances leading to posaconazole underdosing | From posaconazole baseline up to Day100
  A clinical record will be taken twice a week during hospitalization and then once a week to describe clinical symptoms leading to malabsorption: nausea, vomiting, diarrhea, mucositis, colitis. Symptom intensity will be assessed according to the NCI CTCAE v5 classification
Description of circumstances leading to posaconazole underdosing | From posaconazole baseline up to Day100
  Adherence to treatment will be monitored daily during hospitalization by paramedical staff. Once home, adherence will be assessed once a week by the doctor in charge of the patient
Description of circumstances leading to posaconazole underdosing | From posaconazole baseline up to Day100
  All co-medications should be recorded throughout the course of posaconazole treatment, based on data from the patient's medical record
Description of the reasons for administering posaconazole intravenously (IV) | From posaconazole baseline up to Day100
  The physician in charge of the patient should specify the reason(s) for IV administration of the treatment
Description of situations leading to initial non-administration or early discontinuation of posaconazole | From posaconazole baseline up to Day100
  The physician in charge of the patient should specify the situation(s) that led to non-administration or early discontinuation of treatment.
Description of situations leading to initial non-administration or early discontinuation of posaconazole | From posaconazole baseline up to Day 100
  Description of posaconazole-related toxicities according to NCI CTCAE v5 classification
Description of invasive fungal infections occurring | From posaconazole baseline up to 1 year post-transplant and/or through study completion (end of follow-up at the last visit of the last patient included in the study)
  Description of IFI cases according to EORTC classification
Description of patient outcome: incidence of engraftment | Month 1 post-transplant
  Engraftment assessed on hematological reconstitution (number of days of aplasia with PNN <0.5 G/L and platelets < 20, number of platelet and packed cell transfusions)
Description of patient outcome: overall survival (OS) | Up to Day100 and 1 year post-transplant and/or through study completion (end of follow-up at the last visit of the last patient included in the study) or death
  Survival between day 0 of transplantation and date of death or last follow-up
Description of patient outcome: disease-free survival (DFS) | Up to Day100 and 1 year post-transplant and/or through study completion (end of follow-up at the last visit of the last patient included in the study) or documented relapse or death whicvever came first
  Survival between day 0 of transplant and date of relapse, death or last follow-up
Description of patient outcome: non-relapse mortality (NRM) | Up to Day100 and 1 year post-transplant and/or through study completion (end of follow-up at the last visit of the last patient included in the study) or death, whichever came first
  Any death unrelated to relapse or disease progression
Description of patient outcome: incidence of relapse (IR) | Up to Day100 and 1 year post-transplant and/or through study completion (end of follow-up at the last visit of the last patient included in the study) or any documented disease recurrence, whichever came first
  Any documented disease recurrence
Description of patient outcome: cumulative incidence of acute GVHD | Up to Day100 and 1 year post-transplant and/or through study completion (end of follow-up at the last visit of the last patient included in the study)
  Acute GVH grade 2-4 according to Mount Sinai criteria
Description of patient outcome: cumulative incidence of chronic GVHD | Up to Day100 and 1 year post-transplant and/or through study completion (end of follow-up at the last visit of the last patient included in the study)
  Extensive chronic GVH according to NCI criteria
Description of patient outcome: GVHD-free relapse-free survival (GRFS) | Up to Day100 and 1 year post-transplant and/or through study completion (end of follow-up at the last visit of the last patient included in the study) or death
  Median relapse-free survival without grade 3-4 acute GVHD or chronic GVHD requiring systemic treatment
Grade 3 and 4 post-transplant adverse events | Up to Day100 and 1 year post-transplant
  Post-transplant grade 3 and 4 adverse events (dates of occurrence) (NCI CTCAE version 5 criteria)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France, France

IPD SHARING:
Plan to Share IPD: No